CLINICAL TRIAL: NCT05838911
Title: Does Neuromuscular Electrical Stimulation Benefit the Functional Ability of Elderly Patients With Chronic Obstructive Lung Disease
Acronym: NEMS for COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: South Valley University (Other)
Responsible Party: Principal Investigator, Ahmed Samir Abdelkhalik Youssef, lecturer at faculty of physical therapy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BeniSuefU_1
Record Dates: First submitted 2023-04-02; First posted 2023-05-03 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Rehabilitation; Chronic Obstructive Lung Disease; Neuromuscular Electrical Stimulation; Pulmonary Function (FEV1/FVC)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The patients in this group were received the chest physiotherapy program for 20 min each day, for five days a week for three consecutive weeks.
  Interventions: Other: Control Group Chest physical therapy
- Study Group (Experimental): The patients in this group were received the same chest physiotherapy program combined with neuromuscular electrical stimulation (NMES) of gluteus max., quadriceps, and calf muscles performed for 30 min /day for five days a week for three consecutive weeks.
  Interventions: Other: Study Group chest physiotherapy program combined with neuromuscular electrical stimulation (NMES)

INTERVENTIONS:
Other: Study Group chest physiotherapy program combined with neuromuscular electrical stimulation (NMES) — The patients in this group were received the same chest physiotherapy program combined with neuromuscular electrical stimulation of gluteus max., quadriceps, and calf muscles performed for 30 min /day for five days a week for three consecutive weeks.
  Other Names: Chest physical therapy plus NMES
  Arms: Study Group
Other: Control Group Chest physical therapy — The patients in this group were received the chest physiotherapy program for 20 min each day, for five days a week for three consecutive weeks
  Other Names: Chest physical therapy
  Arms: Control Group

SUMMARY:
Background: Patients with COPD often experience skeletal muscle dysfunction. For those who are unable or unwilling to undertake physical training, neuromuscular electrical stimulation (NMES) may provide an alternative method of exercise training.

Objective: To investigate the effects of adding neuromuscular electrical stimulation of gluteus maximus, quadriceps and calf muscles to chest physiotherapy, compared to chest physiotherapy alone, on muscles strength (gluteus max., quadriceps, calf muscles), femoral blood flow physical and pulmonary function in severe COPD Patients.

DETAILED DESCRIPTION:
Material and methods: This study include a group of 60 patients (30 males and 30 females) diagnosed with severe COPD), their age is ranged 65-75 years, they will be randomly divided into two groups; study group (A) 30 patients and study group (B) 30 patients. Study group (A): The patients in this group will receive the chest physiotherapy program for 20 min each day, for five days a week for three consecutive weeks. Study group (B): The patients in this group will receive the same chest physiotherapy program combined with neuromuscular electrical stimulation of gluteus max., quadriceps, calf muscles, performed for 30 min /day for five days a week for three consecutive weeks. Femoral blood Flow, gluteus maximus, quadriceps and calf muscles strength and pulmonary function (FEV1/FVC) will be measured for both groups pre and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD with FEV1/FVC <50% predicted as per the GOLD guidelines.
* Self-reported dyspnea and/or arm fatigue during at least one activity of daily living that required arm exercise.
* Dyspnea and/or physical activity fatigue were self-reported by the Borg Scale.
* Before entering in the study, all patients had their pulmonary function optimized with long-acting bronchodilators and corticosteroids.

Exclusion Criteria:

* • Patients with unstable angina pectoris.

  * Progressive ventricular dysrhythmia.
  * Intermittent claudication.
  * Implanted cardiac pacemakers.
  * Uncontrolled diabetes mellitus.
  * Peripheral vascular disease.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-08-13 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
Six-minute walking test (Physical function assessment | change from baseline to 3 weeks after intervention and 3 days as a follow-up
  The six-minute walking distance (6MWD) was measured according to a standardized protocol.
  * Subjects were instructed to walk at their own pace along a 34.5-m corridor from one end to the other, covering as much ground as possible in the allotted time.
  * Subjects were allowed to stop and rest during the test, but they were instructed to resume walking as soon as they felt able to do
Pulmonary function test | change from baseline to 3 weeks after intervention and 3 days as a follow-up
  Pulmonary capacity and respiratory muscle functions will be assessed using the CPFS/D USB™ 187 Spirometer (Medical Graphics-MGC, St. Paul, MN, USA) with airflow being measured by a 188 calibrated Pitot tube (PreVent, Pneumotach). The participant completed at least three acceptable maximal forced and slow expiratory maneuvers after 15 min the inhalation of 400 mg of salbutamol 190 via a metered-dose inhaler. Forced vital capacity (FVC, L), forced expiratory volume in one second (FEV1, L), FEV1/ FVC, and inspiratory capacity (IC) will be measured according to American Thoracic Society standards
Muscle strength measurement | change from baseline to 3 weeks after intervention and 3 days as a follow-up
  To determine the maximal muscle strength the Lafayette manual muscle test system (USER MANUAL) (MMT) Model 01163, White Plains, New York (10602) of gluteus maximus, quadriceps and calf muscles will be measured on right lower limb.

SECONDARY OUTCOMES:
Blood flow velocimetry measurement | change from baseline to 3 weeks after intervention and 3 days as a follow-up
  To evaluate changes in peripheral perfusion. The standard pulsed-wave Doppler velocimetry of the right femoral artery was performed using sonos 2000 echograph (Philips Envisor )

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim I. I Abu zaid, PhD, Study Director — Department of P.T for internal medicine, Faculty of Physical Therapy, South valley university, Qena, Egypt
Locations (1):
- Department of P.T for internal medicine, Faculty of Physical Therapy, South valley university, Qena, Egypt, Qina, Egypt